CLINICAL TRIAL: NCT06178887
Title: Role of Cardiac Magnetic Resonance Angiography (1.5-T) in the Diagnosis of Cardiac and Thoraco-abdominal Vascular Tree Anomalies in Adult Patients with Turner Syndrome
Brief Title: Role of Cardiac AngioMR in Diagnosis of Cardiac and Vascular Anomalies in Adult Patients with Turner Syndrome
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Vincenzo Rochira, Prof., Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 1001
Record Dates: First submitted 2023-11-27; First posted 2023-12-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Anomaly Heart; Turner Syndrome
MeSH Terms: conditions — Heart Defects, Congenital; Turner Syndrome | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: imaging — cardiac angioMR

SUMMARY:
Considering the high prevalence of cardiovascular disease in Turner syndrome patients, noninvasive cardiac imaging is crucial for diagnosis and follow-up. From the review of the literature, it was evident that the imaging techniques used involved the evaluation of only the thoracic findings, in particular the heart and the thoracic aorta, while no data are currently available on the distal abdominal aorta or iliac arteries, since ultrasound and MRI are interrupted at the diaphragmatic level.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Turner Syndrome
* patients underwent angioMR 1.5 T
* age > 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohort of patients with Turner syndrome > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular and cardiac anomalies | 5 years
  description of the main cardiovascular anomalies found by MRI at the thoracic and abdominal level anomalies in terms of supernumeray arteries and/or veins and measurement of length and diameters of main vascular tracts (e.g. ascending, descending aorta, aortic arch, renal arteries...) or vascular congenital abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Endocrinology of Azienda Ospedaliera-Universitaria di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No